CLINICAL TRIAL: NCT04537403
Title: PET Detection of CCR2 in Human Atherosclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201911199
Record Dates: First submitted 2020-08-17; First posted 2020-09-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aim 1A (Experimental): Normal volunteers and patients with Carotid and Femoral Atherosclerosis who will be having surgery
  Interventions: Drug: Group 1-64CU-DOTA-ECL1i (radioactive imaging medicine)
- Aim 1B (Experimental): Patients with Carotid and Femoral Atherosclerosis who will be managed medically and not having surgery
  Interventions: Drug: Group 2 64CU-DOTA-ECL1i (radioactive imaging medicine)

INTERVENTIONS:
Drug: Group 1-64CU-DOTA-ECL1i (radioactive imaging medicine) — Patients in Group 1, normal volunteers and patients with carotid and femoral artery disease who will be having surgery, will have a 1 day imaging session lasting approximately 60 minutes with an injection of 64CU-DOTA-ECL1i to visualize the carotid and femoral arteries. Patients with carotid and femoral artery disease will have their plaque specimens collected for further sutdy
  Arms: Aim 1A
Drug: Group 2 64CU-DOTA-ECL1i (radioactive imaging medicine) — Patients in Group 2, who are patients with carotid and femoral artery disease who will not be having surgery will have two imaging sessions 7-14 days apart
  Arms: Aim 1B

SUMMARY:
: Use of novel radio-pharmaceutical 64CUDOTA-ECL1i to evaluate arterial atherosclrosis

DETAILED DESCRIPTION:
Using 64CUDOTA-ECL1i to evaluate arterial atherosclrosis in normal volunteers and patients with carotid or femoral arterial atherosclerosis..

ELIGIBILITY:
Inclusion Criteria: Normal Volunteers: 18-40 years of age, non smoker, no history of diabetes, hypertension, or hyperlipidemia. Patients: 50-89 years of age, adequate nutritional status, with or without smoking history, diabetes, hypertension, and hyperlipidema. Both asymptomatic and symptomatic patients with known carotid artery atherosclrosis >70% and scheduled to undergo surgery. Advanced peripheral artery disease.

-

Exclusion Criteria:Inability to receive and sign informed consent. Currently enrolled in another study. Patients who have type 1 diabetes or are in septic shock, receiving steroid therapy, recent history of heavy alcohol consumption, (male >2 drinks per day, and female > 1 drink per day. following extreme diets like Atkins or South Beach diet or with Stage 4 chronic renal failure. Patients with unstable clinical condition that in the opinion of the PI precludes participation in the study. Inability to tolerate 60 minutes in a supine position with arms down at sides. Contraindications to MR imaging, (pacemaker, brain aneurysm clips, shrapnel, etc. Positive pregnancy test or lactating. Have another conditions such as cancer or autoimmune/inflammatory diseases, e.g. rheumatoid arthritis or multiple sclerosis that are known to have increased expression of CCR2.

-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of 64CU-ECL1i , imaging characteristics | 1 or 2 days
  Injecting normal volunteers and patients who have blocked arteries with a single bolus injection. The dose of the injection is 8-10, and the above drug is measured in millicuries, which is a unit of radioactivity.
  the dose of millicuries will be 8-10 millicures

SECONDARY OUTCOMES:
PET/MR camera, imaging performance | 1-2 days
  Utilizing the PET/MR camera using audiography, which can show the presence and size of the blockage

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University CCIR, St Louis, Missouri, United States